CLINICAL TRIAL: NCT01811485
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study to Compare the Effect of 14 Weeks Treatment With LMF237 Bid to Placebo in Patients With Type 2 Diabetes Inadequately Controlled With Vildagliptin 50 mg Bid Monotherapy
Brief Title: Study of Efficacy and Safety LMF237 in Patients With Type 2 Diabetes Mellitus (T2DM) Inadequately Controlled With Vildagliptin Monotherapy
Acronym: CLMF237A1303
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLMF237A1303
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LMF237 50/250 mg (Experimental): Patients took LMF237 50/250 mg twice daily for 14 weeks
  Interventions: Drug: LMF237 50/250 mg; Drug: LMF237 50/500 mg
- LMF237 50/500 mg (Experimental): Patients took LMF237 50/500 mg (with a starting dose of LMF 237 50/250 mg for 2 weeks) twice daily for 14 weeks
  Interventions: Drug: LMF237 50/250 mg
- Placebo (Placebo Comparator): Patients took matching placebo of LMF237 (vildagliptin 50 mg) twice daily for 14 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LMF237 50/250 mg — Corresponds to vildagliptin 50 mg twice daily and metformin 250 mg twice daily
  Arms: LMF237 50/250 mg; LMF237 50/500 mg
Drug: LMF237 50/500 mg — Corresponds to vildagliptin 50 mg twice daily and metformin 500 mg twice daily
  Arms: LMF237 50/250 mg
Drug: Placebo — Matching placebo of LMF237 (contained vildagliptin 50 mg as active ingredient) twice daily
  Arms: Placebo

SUMMARY:
The purpose of the study was to evaluate the efficacy and safety of LMF237 50/250 mg and 50/500 mg bid in Japanese patients with T2DM inadequately controlled with vildagliptin monotherapy. This study was conducted to support registration of the fixed-dose combination of vildagliptin and metformin for the treatment of T2DM in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes inadequately controlled with diet, exercise and oral anti-diabetic therapy
* HbA1c in the range of 7.0-10.0%
* Body mass index in the range of 20-35 kg/m^2

Exclusion Criteria:

* Type 1 diabetes, monogenic diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes
* Significant heart diseases Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- Japan (23):
  - Novartis Investigative Site, Chikushino-shi, Fukuoka
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Koga, Ibaraki
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yatsushiro, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Ageo, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Katsushika-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Nerima-ku, Tokyo
  - Novartis Investigative Site, Shibuya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LMF237 50/250 mg | LMF237 50/500 mg | Placebo
Started | 56 ("Started" indicates randomized patients) | 59 | 56
Completed | 54 | 55 | 51
Not Completed | 2 | 4 | 5
Not completed — Adverse Event | 1 | 3 | 2
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 3
Not completed — Administrative problems | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set
Groups:
- Total: Total of all reporting groups
Arm/Group | LMF237 50/250 mg | LMF237 50/500 mg | Placebo | Total
Number analyzed (Participants) | 56 | 59 | 56 | 171
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (11.24) | 58.3 (10.50) | 56.2 (9.75) | 57.0 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 16 | 49
  Male | 41 | 41 | 40 | 122

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at 14 Weeks Between Treatment Groups
Description: HbA1c was performed on a blood sample obtained and measured by High performance liquid chromatography (HPLC). HPCL was performed at a central laboratory.
Time Frame: Baseline to 14 weeks
Population: Full analysis set consisted of all randomized patients who received at least one dose of study medication and had at least one post-randomization efficacy parameter measurement.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Groups:
- Pooled LMF237: All patients who took LMF237 50/250 mg or LMF237 50/500 mg twice daily for 14 weeks were pooled together as reporting group.
Arm/Group | Pooled LMF237 | Placebo
Number analyzed (Participants) | 115 | 56
percentage of glycosylated haemoglobin | -0.83 (0.06) | 0.14 (0.08)

2. Secondary Outcome: Change From Baseline in HbA1c at 14 Weeks Within LMF237 Treatment Groups
Description: HbA1c will be performed on a blood sample obtained and measured by HPLC. HPCL was performed at a central laboratory.
Time Frame: Baseline to 14 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | LMF237 50/250 mg | LMF237 50/500 mg
Number analyzed (Participants) | 56 | 59
percentage of glycosylated haemoglobin | -0.61 (0.06) | -1.04 (0.06)

3. Secondary Outcome: Percentage of Patients Meeting Responder Rates in HbA1c
Description: Responder rate was analyzed in categories: 1. Endpoint HbA1c ≤ 6.5% 2. Endpoint HbA1c < 7% 3. Endpoint HbA1c < 7% in patients with baseline HbA1c ≤ 8% 4. Endpoint HbA1c < 6.9% 5. HbA1c reduction from baseline at endpoint ≥ 1% 6. HbA1c reduction from baseline at endpoint ≥ 0.5%.
  Categories 1, 2, and 4 - 'n' includes only patients with baseline HbA1c > 6.5%, ≥ 7%, ≥ 6.9% and endpoint HbA1c measurement. Category 3, 'n' includes only patients with 7% ≤ baseline HbA1c ≤ 8% and endpoint HbA1c. Category 5 and 6, 'n' indicates number of patients with both baseline and endpoint HbA1c measurements.
Time Frame: Baseline, 14 weeks
Population: The full analysis set (FAS) consisted of all randomized patients who received at least one dose of study medication and had at least one post-randomization efficacy parameter measurement.
Measure: Number; unit: Percentage of patients
Arm/Group | Pooled LMF237 | Placebo
Number analyzed (Participants) | 115 | 56
Percentage of patients
  HbA1c ≤ 6.5% (n=115, 56) | 27.8 | 0.0
  HbA1c < 7.0% (n= 107, 52) | 45.8 | 13.5
  HbA1c < 7.0% with baseline HbA1c ≤ 8.0% (n=69,33) | 66.7 | 18.2
  HbA1c < 6.9% (n= 111, 54) | 45.0 | 9.3
  Reduction of HbA1c ≥ 1% (n= 115, 56) | 36.5 | 1.8
  Reduction of HbA1c ≥ 0.5% (n= 115, 56) | 73.9 | 16.1

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at 14 Weeks
Description: FPG was performed on a blood sample obtained and analyzed at a central laboratory.
Time Frame: Baseline to 14 weeks
Population: FAS consisted of all randomized patients who received at least one dose of study medication and had at least one post-randomization efficacy parameter measurement.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pooled LMF237 | Placebo
Number analyzed (Participants) | 115 | 56
mg/dL | -13.02 (2.83) | 16.54 (4.06)

5. Secondary Outcome: Number of Patients With Adverse Events (Including Hypoglycemia), Serious Adverse Events and Death
Description: The occurrence of adverse events were sought by non-directive questioning of the patient at each visit. Adverse events are defined as appearance or worsening of any undesirable symptom, sign (including an abnormal laboratory finding), or medical conditions. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: 14 weeks
Population: Safety set (SAF): consists of all patients who received at least one dose of study medication.
Measure: Number; unit: Patients
Arm/Group | LMF237 50/250 mg | LMF237 50/500 mg | Placebo
Number analyzed (Participants) | 56 | 59 | 56
Patients
  Any AE (Serious and non-serious) | 25 | 25 | 38
  Serious AEs | 0 | 1 | 2
  Death | 0 | 0 | 0

ADVERSE EVENTS:
Description: Safety set (SAF): The SAF consists of all patients who received at least one dose of study medication.
Groups:
- POOLED LMF237: All patients who has received LMF237
- LMF237 50/250mg: Patients took LMF237 50/250 mg twice daily for 14 weeks
- LMF237 50/500mg: Patients took LMF237 50/500 mg (with a starting dose of LMF 237 50/250 mg for 2 weeks) twice daily for 14 weeks
Arm/Group | POOLED LMF237 | LMF237 50/250mg | LMF237 50/500mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/115 | 0/56 | 1/59 | 2/56
Other Adverse Events (participants affected / at risk) | 22/115 | 7/56 | 15/59 | 17/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | POOLED LMF237 (N=115) | LMF237 50/250mg (N=56) | LMF237 50/500mg (N=59) | Placebo (N=56)
Epiglottitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | POOLED LMF237 (N=115) | LMF237 50/250mg (N=56) | LMF237 50/500mg (N=59) | Placebo (N=56)
Constipation (Gastrointestinal disorders) | 3 | 0 | 3 | 0
Gastritis (Gastrointestinal disorders) | 2 | 2 | 0 | 3
Nausea (Gastrointestinal disorders) | 6 | 1 | 5 | 2
Asthenia (General disorders) | 3 | 0 | 3 | 1
Nasopharyngitis (Infections and infestations) | 11 | 4 | 7 | 10
Lipase increased (Investigations) | 0 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 3 | 0 | 3 | 0
Tremor (Nervous system disorders) | 3 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.